CLINICAL TRIAL: NCT05892705
Title: Can Subarachnoid Dexmedetomidine Decrease the Incidence of Postoperative Nausea and Vomiting and Shivering With Minimal Hemodynamic Instability in CS?
Brief Title: Intrathecal Dexmedetomidine to Decrease Postoperative Nausea and Vomiting and Shivering.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Shaimaa Mohamed Samir Ezzat Rakhia, MD, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: FAMSU R 120 / 2021
Record Dates: First submitted 2023-05-14; First posted 2023-06-07 (Actual); Last update posted 2023-06-07 (Actual); Status verified 2023-05

CONDITIONS: Intrathecal Dexmedetomidine
MeSH Terms: interventions — Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Study drug (dexmedetomidine intrathecal) (Active Comparator): 5 mcg dexmedetomidine intrathecally injected with 10 mg hyperbaric bupivacaine during spinal anesthesia for caesarean section.
  Interventions: Drug: Dexmedetomidine Injection [Precedex]
- Control (saline) (Placebo Comparator): 0.2 ml normal saline intrathecally injected with 10 mg hyperbaric bupivacaine during spinal anesthesia for caesarean section.
  Interventions: Drug: Dexmedetomidine Injection [Precedex]

INTERVENTIONS:
Drug: Dexmedetomidine Injection [Precedex] — intrathecal injection of 5 mcg dexmedetomidine

SUMMARY:
Background: Highly selective α-2 agonist dexmedetomidine in increasingly used as an intrathecal adjuvant for caesarean section performed under subarachnoid block.

Aim of the Study: The aim of the study is to determine whether low dose dexmedetomidine added to local anesthetic for spinal anesthesia will attenuate perioperative nausea and vomiting and shivering in lower segment caesarean section (LSCS) with minimal hemodynamic instability or not.

Patients and Methods: Sixty parturients planned for elective CSs under spinal anesthesia were enrolled in this prospective controlled study and randomly divided into two equal groups. Spinal block was achieved with 10mg hyperbaric bupivacaine 0.5% plus 5µg dexmedetomidine (group D) (dexmedetomidine group) or 0.2 ml normal saline (group C) (control group). Hemodynamic parameters, incidence of nausea and vomiting and shivering were recorded.

Keywords: Dexmedetomidine, Cesarean Section, Bupivacaine, Spinal Anesthesia, Shivering, PONV

ELIGIBILITY:
Inclusion Criteria:

* Medically free pregnant Female from 18 to 30 yrs old.
* Undergoing elective LSCS.
* Body mass index less than 40.
* Consenting for sub arachnoid anesthesia.
* Coagulation profile is within normal ranges.

Exclusion Criteria:

* Emergency LSCS.
* Patient refusal enrollment in the study.
* Allergy to the medications.
* Coagulopathy or anticoagulation drugs.
* Fetal or Maternal comorbidities.

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2023-01-15 (Actual); Study Completion 2023-01-15 (Actual)

PRIMARY OUTCOMES:
Effect of subarachnoid dexmedetomidine on hemodynamic parameters. | Two hours
  Measure heart rate, blood pressure, temperature, oxygen saturation

SECONDARY OUTCOMES:
Effect of subarachnoid dexmedetomidine on incidence of postoperative nausea and vomiting (PONV) and shivering. | Six hours
  Note occurrence of postoperative nausea or vomiting and note occurrence of shivering and measure the degree.

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University, Cairo, Abbasia, Egypt

IPD SHARING:
Plan to Share IPD: No